CLINICAL TRIAL: NCT06164080
Title: The Effect Of Antenatal Corticosteroids On Early And Late Perinatal Outcomes In Late Preterm Pregnant Women
Brief Title: The Effect Of Antenatal Corticosteroids On Early And Late Perinatal Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2011-KAEK-25 2021/05-10
Record Dates: First submitted 2023-04-04; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Preterm Pregnancy; Antenatal Corticosteroid; Perinatal Problems
Keywords: Antenatal corticosteroids; Late preterm pregnancy; Late perinatal outcomes
MeSH Terms: interventions — Betamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antenatal corticosteroid non-administration (No Intervention): Pregnant women who did not use antenatal corticosteroid before 34 weeks
- Antenatal corticosteroid administration (Active Comparator): Pregnant women using antenatal corticosteroids for any reason before 34 weeks
  Interventions: Other: participants receiving Corticosteroid

INTERVENTIONS:
Other: participants receiving Corticosteroid — Pregnant women using antenatal corticosteroids for any reason before 34 weeks
  Other Names: betamethasone; dekort
  Arms: Antenatal corticosteroid administration

SUMMARY:
In this study, the investigators aims to evaluate whether antenatal corticosteroid administration to women likely to give birth in the late preterm period will reduce early and late neonatal complications and contribute to the literature in this sense.

DETAILED DESCRIPTION:
This study is a single-center prospective case-control study investigating the effect of antenatal corticosteroids administered in the late preterm period on early and late perinatal outcomes. 459 patients who gave birth between 34-37 weeks between June 1,2021 to October 1,2022 in the Obstetrics and Gynecology Clinic of the University of Health Sciences were included. Patient were divided into two groups antenatal corticosteroid administration (n:231) and non-administration (n:228). Postpartum early and late perinatal outcomes were compared between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who had normal vaginal delivery, cesarean section or operative delivery between 34-37 weeks
* Singleton pregnancies resulting in a live birth

Exclusion Criteria:

* Twin pregnancies
* All births before 34 weeks or after 37 weeks
* Pregnant women with intrauterine ex fetus
* Fetuses with major congenital and chromosomal abnormalities
* Pregnant women who administrated antenatal corticosteroids for any reason before 34 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 459 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
The results of antenatal corticosteroid effects | 16 months
  intramuscular 3 mg betamethasone (dekort 8mg/2 ml) corticosteroid injection in perinatal period

SECONDARY OUTCOMES:
Other consequences of antenatal corticosteroid effects in late term pregnant women | 16 months
  Other consequences of antenatal corticosteroid administered in late preterm pregnant women in the neonatal period are the need for neonatal intensive care due to reasons other than respiratory distress, respiratory complications such as pneumonia, other complications such as sepsis, perinatal death, chronic lung disease (even after 28 days of birth, oxygen need) long-term outcomes in postnatal infants ( third month, sixth month, twelfth month, emotional and emotional consequences in the family, and maternal side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Bursa, Turkey (Türkiye)